CLINICAL TRIAL: NCT05144802
Title: Accuracy of Dexcom G6® and FreeStyle Libre® Sensors in Standardized Hypoxemia Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FOX
Record Dates: First submitted 2021-10-29; First posted 2021-12-03 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: CGM (Continuous Glucose Monitoring)
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 : FreeStyle Libre 2 on right arm and Dexcom G6 on left arm (Experimental): In this group, participants will be continuously monitored for their interstitial glucose level with 2 CGM devices : FreeStyle Libre 2 will be applied on right arm and Dexcom G6 will be applied on left arm.
  Interventions: Procedure: acute hypoxia
- group 2 : 2 FreeStyle Libre 2 on left arm and Dexcom G6 on right arm (Active Comparator): In this group, participants will be continuously monitored for their interstitial glucose level with 2 CGM devices : Dexcom G6 will be applied on right arm and FreeStyle Libre 2 will be applied on left arm.
  Interventions: Procedure: acute hypoxia

INTERVENTIONS:
Procedure: acute hypoxia — Participants will be exposed to a 3-hour acute hypoxia

SUMMARY:
The major aim is to evaluate accuracy of 2 Continuous Glucose Monitoring Systems (CGMS) : Dexcom G6® and FreeStyle Libre® in standardized hypoxemia conditions (artificial normobaric hypoxia).

Our purpose is to demonstrate the good performance and calibration of these CGM sensors in hypoxemia conditions.

ELIGIBILITY:
Inclusion Criteria: all population

* No history of respiratory diseases (childhood asthma, respiratory allergies, exercise-induced asthma or dyspnea)
* Willing to participate and able to sign an informed consent form (ICF)
* Being affiliated with the French Social Security

Inclusion Criteria:Patients with diabetes

* type 1 diabetes mellitus or type 2 diabetes mellitus (ADA definition)
* Age : 18 to 75 years
* stable diabetes treatment for more than 3 months
* no diabetic retinopathy
* no diabetic neuropathy
* no cardiovascular diseases
* no contra-indication for coronary computed tomography angiography or myocardial perfusion scintigraphy.

Inclusion Criteria: Healthy volunteers

* Age : 18 ; 40 years
* No diabetes
* No persistant drug use > 3 months except contraception
* Body mass index : [18,5 - 29,9] kg/m2

Non-inclusion criteria : all population

* Active smokers
* Pregnant or breastfeeding women, women of childbearing age without effective contraception
* Known allergies to the patch.
* Skin lesions at the sensor site that may interfere with sensor placement or accuracy
* Major cardiovascular complications within the past 3 months
* Decompensated congestive heart failure
* Chronic respiratory failure
* Chronic renal failure
* Resting ambient air O2 saturation ≤95%.
* Treatment with systemic corticosteroids
* Severe hypertension (≥180 mmHg systolic pressure or ≥ 100 mmHg diastolic pressure)
* Any concomitant disease or condition that the investigator believes may compromise patient safety or affect the conduct of the study
* Anemia (Hb<12g/dl)
* History of severe mountain sickness
* Concurrent participation in another clinical research study,
* Persons benefiting from enhanced protection

Non-inclusion criteria: Patients with diabetes

* Absolute contraindications to physical activity (HAS definitin) :
* Pulmonary arterial hypertension (> 60 mm Hg)
* Presence of intra-cardiac thrombus
* Acute pericardial effusion
* Severe obstructive cardiomyopathy
* Symptomatic aortic stenosis
* Recent thrombophlebitis with or without pulmonary embolism

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Assess accuracy of interstitial glucose values measured respectively by FreeStyle® Libre and Dexcom® G6 compared to blood glucose values in standardized hypoxemia conditions in patients with diabetes and in healthy volunteers. | Day 1
  Mean absolute relative difference (MARD)

SECONDARY OUTCOMES:
Safety of acute hypoxia | Day 1
  Arterial blood oxygen saturation (Sp02)
Tolerability of acute hypoxia | Day 1
  Lake Louise Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Poitiers, France